CLINICAL TRIAL: NCT00699192
Title: A Multicenter, Double-blind, Randomized, Parallel-group Study to Evaluate the Safety, Tolerability, and Efficacy of Once Daily Amlodipine/Valsartan 5/80 mg as Compared to Amlodipine/Valsartan 5/40 mg or to Amlodipine 5 mg Once Daily in Elderly Patients With Essential Hypertension Not Adequately Controlled After Four Weeks on Amlodipine 5 mg Once Daily
Brief Title: Safety, Tolerability, and Efficacy of Once Daily Amlodipine/Valsartan 5/80 as Compared to Amlodipine/Valsartan 5/40 or to Amlodipine 5 mg Monotherapy in Patients 65 Years of Age and Older With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAA489A2318
Record Dates: First submitted 2008-06-09; First posted 2008-06-17 (Estimated); Results first posted 2011-06-06 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension
Keywords: Blood pressure; hypertension; elderly
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Amlodipine/Valsartan 5/80 mg (Experimental): 1 capsule amlodipine 5 mg, 1 capsule valsartan 80 mg once daily
  Interventions: Drug: Amlodipine 5 mg; Drug: Valsartan 80 mg
- Amlodipine/Valsartan 5/40 mg (Active Comparator): 1 capsule amlodipine 5 mg, 1 capsule valsartan 40 mg once daily
  Interventions: Drug: Amlodipine 5 mg; Drug: Valsartan 40 mg
- Amlodipine 5 mg (Active Comparator): 1 capsule amlodipine 5 mg, 1 capsule placebo to match valsartan once daily
  Interventions: Drug: Amlodipine 5 mg; Drug: Placebo

INTERVENTIONS:
Drug: Amlodipine 5 mg — 1 capsule amlodipine 5 mg orally once daily
Drug: Valsartan 80 mg — 1 capsule valsartan 80 mg orally once daily
  Arms: Amlodipine/Valsartan 5/80 mg
Drug: Valsartan 40 mg — 1 capsule valsartan 40 mg orally once daily
  Arms: Amlodipine/Valsartan 5/40 mg
Drug: Placebo — 1 capsule placebo to match valsartan orally once daily
  Arms: Amlodipine 5 mg

SUMMARY:
To characterize the safety, tolerability, and efficacy profile of amlodipine/valsartan 5/80 mg as compared to amlodipine/valsartan 5/40 mg (with optional titration to 5/80 mg) and amlodipine 5 mg monotherapy in elderly patients (≥ 65 years of age) with essential hypertension. All three regimens are expected to be well tolerated.

ELIGIBILITY:
Inclusion criteria

* Provide written informed consent before any assessment was performed.
* Male or female at least 65 years of age.
* Diagnosed as having hypertension:

  * At Visit 1/Screening, treatment naïve patients had to have a mean seated SBP ≥ 155 mmHg and < 180 mmHg; patients undergoing washout from their previous antihypertension medication had to have a mean seated SBP <180 mmHg.
  * At Visit 2/Single-blind run-in entry, all patients had to have a mean seated SBP ≥ 155 mmHg and < 180 mmHg.
  * At Visit 3/Core double-blind treatment period entry, all patients had to have a mean seated SBP ≥ 145 mmHg and < 180 mmHg.
* Ability to communicate and comply with all study requirements including measuring their blood pressure at home, daily as instructed, using the home blood pressure monitor provided by the Sponsor.
* Female patients had to be post-menopausal for at least one year.

Exclusion criteria

* Severe hypertension (mean seated SBP ≥ 180 mmHg and/or a mean seated DBP ≥ 110 mmHg).
* History of secondary hypertension (including primary aldosteronism, renovascular hypertension, pheochromocytoma, etc.).
* Use of three or more antihypertensive drugs. Dual fixed dose combination therapy was considered as two antihypertensive drugs.
* Administration of any agent indicated for the treatment of hypertension after Visit 1, with the permitted exception of those antihypertensive medications requiring tapering down (e.g. beta-blocker and/or clonidine) commencing with Visit 1.
* Known moderate or malignant retinopathy. Moderate was defined as retinal signs of hemorrhage, microaneurysm, cotton-wool spot, hard exudates, or a combination thereof; malignant defined as signs of moderate retinopathy plus swelling of the optic disk.
* Known or suspected contraindications, including history of allergy or hypersensitivity to angiotensin receptor blockers (ARB), calcium channel blockers (CCB), or to drugs with similar chemical structures.
* History of cerebrovascular accident, thrombotic stroke, or transient ischemic attack.
* Significant history of coronary artery disease (CAD) such as any history of myocardial infarction (MI), angina pectoris, and all types of revascularization procedures.
* History of or diagnosis of congestive heart failure Grade II-IV according to the New York Heart Association (NYHA) classification.
* Clinically significant valvular heart disease.
* All patients with Type 1 diabetes mellitus and those patients with Type 2 diabetes mellitus who, in the opinion of the investigator, were not well controlled. Patients who needed oral anti-diabetic medication to adequately control their Type 2 diabetes had to be on a stable dose of oral anti-diabetic medication for at least 4 weeks prior to Visit 1.
* Concomitant potentially life threatening arrhythmia or symptomatic arrhythmia.
* Second or third degree heart block with or without a pacemaker.
* Significant hepatic disease, as demonstrated by any one of the following: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values greater than two times the upper limit of normal at Visit 1, a history of hepatic encephalopathy, a history of esophageal varices, or a history of a portocaval shunt.
* Evidence of renal impairment as determined by any one of the following: glomerular filtration rate (GFR) < 50 ml/min/1.73m2 as measured by the Modification of Diet in Renal Disease (MDRD) formula at Visit 1, a history of dialysis, or a history of nephrotic syndrome.
* History of clinically significant allergies including asthma and/or multiple drug allergies.
* Any surgical or medical condition with the potential to significantly alter the absorption, distribution, metabolism, or excretion of any drug including but not limited to any of the following: history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling, or gastric banding, currently active or inactive inflammatory bowel syndrome within 12 months prior to Visit 1, currently active gastritis, ulcers, or gastrointestinal/rectal bleeding, or urinary tract obstruction regarded as clinically meaningful by the investigator.
* Any condition, not identified in the protocol, that, in the opinion of the investigator or the Novartis monitor, placed the patient at higher risk from his/her participation in the study, or was likely to prevent the patient from complying with the requirement of the study or completing the trial period.
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there was evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
* Any chronic inflammatory condition needing chronic anti-inflammatory therapy.
* History of drug or alcohol abuse within the last 2 years.
* Use of investigational drugs at the time of enrollment, or within 30 days prior to Visit 1 (Week 8).
* Inability to communicate and comply with all study requirements including the unwillingness or inability to provide informed consent.
* Persons directly involved in the execution of this protocol.
* History of non-compliance to medical regimens, or patients unwilling to comply with the study protocol.
* Any severe, life-threatening disease within the past five years.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 965 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Czechia (6):
  - Novartis Investigative site, Brno
  - Investigative site Czech Republic, Chrudim
  - Investigative sites Czech Repbulic, Hodonín
  - Investigative site Czech Repbulic, Jičín
  - Sites in Czech Republic, Náchod
  - Investigative sites Czech Republic, Prague
- Finland (4):
  - Investigative site Finland, Helsinki
  - Investigative site Finland, Joensuu
  - Investigative site Finland, Kerava
  - Investigative site Finland, Tampere
- Investigative site France, Paris, France
- Investigative site Germany, Berlin, Germany
- Investigative site Hungary, Budapest, Hungary
- Investigative site Italy, Rome, Italy
- Investigative site Poland, Warsaw, Poland
- Investigative site Slovakia, Bratislava, Slovakia
- Investigative site Spain, Valencia, Spain
- Investigative site Sweden, Malmo, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 965 patients were enrolled in the study. Of these, 819 met the criteria for entry into the double-blind phase of the study where efficacy and safety were evaluated.
Period: Overall Study
Arm/Group | Amlodipine/Valsartan 5/80 mg | Amlodipine/Valsartan 5/40 mg | Amlodipine 5 mg
Started | 275 | 272 | 272
Completed | 259 | 260 | 261
Not Completed | 16 | 12 | 11
Not completed — Missing | 1 | 1 | 1
Not completed — Adverse Event | 9 | 4 | 3
Not completed — Abnormal test procedure result(s) | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 4
Not completed — Administrative problems | 1 | 3 | 1
Not completed — Protocol Violation | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amlodipine/Valsartan 5/80 mg | Amlodipine/Valsartan 5/40 mg | Amlodipine 5 mg | Total
Number analyzed (Participants) | 275 | 272 | 272 | 819
Age Continuous [Mean (Standard Deviation); unit: years] | 71.8 (5.01) | 71.6 (5.38) | 71.4 (5.44) | 71.6 (5.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 138 | 142 | 432
  Male | 123 | 134 | 130 | 387

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Baseline to End of Study (Week 8)
Description: At study entry, blood pressure (BP) was measured in both arms with an automatic BP monitor. The arm with the higher systolic BP reading was used for all measurements throughout the study. At each study visit, 3 separate sitting BPs were obtained 23-26 hours post-dose with at least 2 minutes between measurements and with the cuff fully deflated. Mean BP was automatically calculated from the 3 readings. A negative change from baseline indicates lowered BP.
Time Frame: Baseline to end of study (Week 8)
Population: The Full Analysis Set (FAS) population: All randomized patients who had a baseline and at least one post-baseline assessment an efficacy variable. For the subjects who did not complete the Week 8 assessments, an LOCF (last observation carried forward) approach was used.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine/Valsartan 5/80 mg | Amlodipine/Valsartan 5/40 mg | Amlodipine 5 mg
Number analyzed (Participants) | 272 | 269 | 268
mmHg | -11.1 (12.68) | -12.3 (13.23) | -6.9 (14.00)

2. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to End of Study (Week 8)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine/Valsartan 5/80 mg | Amlodipine/Valsartan 5/40 mg | Amlodipine 5 mg
Number analyzed (Participants) | 272 | 269 | 268
mmHg | -4.2 (8.04) | -5.3 (8.19) | -1.7 (7.26)

3. Secondary Outcome: Percentage of Patients Achieving a Systolic Blood Pressure Response at Week 8
Description: A systolic blood pressure response was defined as a msSBP < 140 mmHg or ≥ 15 mmHg reduction from baseline at the end of the study (Week 8). At study entry, blood pressure (BP) was measured in both arms with an automatic BP monitor. The arm with the higher systolic BP reading was used for all measurements throughout the study. At each study visit, 3 separate sitting BPs were obtained 23-26 hours post-dose with at least 2 minutes between measurements and with the cuff fully deflated. Mean BP was automatically calculated from the 3 readings.
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Amlodipine/Valsartan 5/80 mg | Amlodipine/Valsartan 5/40 mg | Amlodipine 5 mg
Number analyzed (Participants) | 272 | 269 | 268
Percentage of patients | 46.0 | 48.3 | 34.0

4. Secondary Outcome: Percentage of Patients Achieving Systolic Blood Pressure Control at the End of the Study (Week 8)
Description: Systolic blood pressure control was defined as a msSBP < 140 mmHg at the end of the study (Week 8). At study entry, blood pressure (BP) was measured in both arms with an automatic BP monitor. The arm with the higher systolic BP reading was used for all measurements throughout the study. At each study visit, 3 separate sitting BPs were obtained 23-26 hours post-dose with at least 2 minutes between measurements and with the cuff fully deflated. Mean BP was automatically calculated from the 3 readings.
Time Frame: End of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Amlodipine/Valsartan 5/80 mg | Amlodipine/Valsartan 5/40 mg | Amlodipine 5 mg
Number analyzed (Participants) | 272 | 269 | 268
Percentage of patients | 31.3 | 37.5 | 20.5

5. Secondary Outcome: Percentage of Patients Achieving Overall Blood Pressure Control at the End of the Study (Week 8)
Description: Overall blood pressure control was defined as a msSBP < 140 mmHg and msDBP < 90 mmHg at the end of the study (Week 8). At study entry, blood pressure (BP) was measured in both arms with an automatic BP monitor. The arm with the higher systolic BP reading was used for all measurements throughout the study. At each study visit, 3 separate sitting BPs were obtained 23-26 hours post-dose with at least 2 minutes between measurements and with the cuff fully deflated. Mean BP was automatically calculated from the 3 readings.
Time Frame: End of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Amlodipine/Valsartan 5/80 mg | Amlodipine/Valsartan 5/40 mg | Amlodipine 5 mg
Number analyzed (Participants) | 272 | 269 | 268
Percentage of patients | 30.9 | 36.4 | 19.0

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Adverse events (AE) could be volunteered by the subject, discovered during general questioning by the investigator, or detected through physical examination, laboratory test, or other means. Medical conditions/diseases present before starting study treatment were only considered AEs if they worsened after starting study treatment.
Arm/Group | Amlodipine/Valsartan 5/80 mg | Amlodipine/Valsartan 5/40 mg | Amlodipine 5 mg
Serious Adverse Events (participants affected / at risk) | 5/274 | 2/272 | 1/272
Other Adverse Events (participants affected / at risk) | 0/274 | 0/272 | 0/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine/Valsartan 5/80 mg (N=274) | Amlodipine/Valsartan 5/40 mg (N=272) | Amlodipine 5 mg (N=272)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Ophthalmoplegia (Eye disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.